CLINICAL TRIAL: NCT04149314
Title: PGDT With the "Hypotension Prediction Index" to Reduce the Number and Duration of Intraoperative Hypotension and the Incidence of Renal Failure in Patients Undergoing Lung Surgery
Brief Title: The "Hypotension Prediction Index" in Patients Undergoing Lung Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPI III
Record Dates: First submitted 2019-07-22; First posted 2019-11-04 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Hypotension; Hemodynamic Instability; Renal Failure; Myocardial Injury; Anesthesia
Keywords: HPI; Thoracic Surgery; Single-Lung ventilation
MeSH Terms: conditions — Hypotension; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: The study is designed as a single center randomized prospective blinded interventional trial comparing goal directed hemodynamic management using HPI compared to standard care.
Who Masked: Investigator
Masking Description: In the interventional study group HPI monitoring is used for hemodynamic optimization while in the control group HPI monitoring is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): Interventional group (hemodynamic optimization based on HPI).
  Interventions: Other: HPI based hemodynamic optimization algorithm
- Control (No Intervention): Control group (blinded HPI monitoring, standard anesthesia care).

INTERVENTIONS:
Other: HPI based hemodynamic optimization algorithm — Interventional patients will be treated by a HPI-based hemodynamic optimization protocol including HPI, Stroke volume, cardiac index and mean arterial pressure.
  Arms: Interventional

SUMMARY:
The "Hypotension Prediction Index (HPI)" was established by the Edwards Lifescience Company (Irvine, California, USA) and is CE certified. As part of the Edwards Acumen Decision-Support-Software-Suite the HPI is supported by the minimal invasive FloTrac Sensor. The HPI displays the probability of an occurring hypotension. The software was established with the help of 20.000 analyzed patient events. If the upper limit of the HPI is reached, the software is alarming the treating physician 8. At the university hospital of Giessen HPI analyses are used in the daily clinical routine as well as for scientific purposes. Preliminary data of the HPI-I-Trial ("Influence of the Hypotension Prediction Index on the number and duration of intraoperative hypotension in primary hip-endoprothetic replacement", University Hospital of Giessen) included patients, which underwent hip-endoprothetic replacement surgery and revealed that the use of HPI with a goal directed therapy (GDT) protocol compared to standard care significantly reduced the incidence and duration of intraoperative hypotension. Therefore HPI with GDT might reduce the incidence of hypotension related complications in a sicker patient cohort.

The aim of the study is to investigate whether a goal directed treatment according to the Hypotension Prediction Index compared to standard care can reduce the incidence of intraoperative hypotension in patients under single lung ventilation.

DETAILED DESCRIPTION:
Monitoring of blood pressure is a basic tool to assess the patients' hemodynamic status. Physiological blood pressure is usually close to 120/80 mmHg. Hypotension is not clearly defined as shown in previous studies 1, 20, 21. Some studies defined hypotension as a systolic blood pressure below 100 mmHg or a mean arterial pressure below 60 mmHg 1,2. Depending on the definition intraoperative hypotension (IOH) hypotension can occur in 38% of patients undergoing non-cardiac surgery. 53% of these patients die within one year. Monk et al. noted that the 1-year-mortality was raised by 3.6% for every minute the systolic blood pressure was below 80 mmHg. The risk of mortality was raised up to 1.4 times when the MAP was under 55 mmHg for more than 10 minutes 3. Additionally, in 2015 it was shown that even short duration of MAP under 55 mmHg is associated with a high risk for acute kidney injury and myocardial infarction 4. A recent definition of hypotension was published by of Vernooij et al. that defined IOH as a decrease of MAP < 65 mmHg for more than one minute in this study 22. Perioperative hypotension is a complication that can occur in the induction period and in the following phase. Recent unpublished data from the Sessler group presented at the 2018 ASA meeting in San Francisco showed that about 1/3 of hypotensive episodes are unrelated to surgery as those occur before the surgeon is in the OR 28. The reasons for hypotension can be found in vasodilatation (e. g. drug induced), volume deficit (based on blood loss), or negative inotropic effect of surgery and anesthetic drugs (reduced left ventricular function). Main factors causing intraoperative hypotension according to literature are age, preexisting diseases (especially ASA > 3), duration of surgery, acuteness of surgery (emergency), anti-hypertensive medication and anesthesia combining general and regional anesthesia 5,6. Complications related to hypotension can be detected in most organ systems. One important source of hypotension-associated complications are cardiovascular complications. Recently, a syndrome that was termed myocardial injury after non-cardiac surgery (MINS) was shown to be associated with hypotension and lead to increased postoperative mortality rate 23, 24. Acute kidney injury (AKI) affects up to 25% of patients in the intensive care unit 7. Liu et al. described that an episode of relative hypotension is often followed by AKI (a decrease in systolic blood pressure relative to pre-morbid value was a significant independent predictor of the development of AKI and of RIFLE classes I and F; odds ratio 1.084 for every -1 mmHg change in systolic blood pressure) 8. As stated, 'normotensive renal failure' is not common and a rare phenomenon in the absence of septic and other complications. This results are supported by other publications, like Lehmann et al. 9. Their results indicate that the risk of AKI was related to the severity of hypotension with an odds ratio (OR) of 1.03, 95% CI 1.02-1.04 (p < 0.0001) per 1 mmHg decrease in minimum MAP ≥ 80 mmHg. For each additional hour MAP was less than 70, 60, 50 mmHg, the risk of AKI increased by 2% (OR 1.02, 95% CI 1.00-1.03, p = 0.0034), 5% (OR 1.05, 95% CI 1.02-1.08, p = 0.0028), and 22% (OR 1.22, 95% CI 1.04-1.43, p = 0.0122).

Renal failure poses a relevant complication in the perioperative phase 5, 6. Over the last decade the cell cycle arrest biomarkers TIMP-2- and IGFBP7-quantification (Nephrocheck) has been successfully evaluated for the detection of AKI 7. The main advantage of both parameters is the opportunity of early detection of AKI and its point-of-care design, which makes them especially for the use on the intensive care unit valuable. Based on these facts, the predictive measurement of blood pressure is of great interest for the anesthesiologist to optimize patients' postoperative outcome.

The "Hypotension Prediction Index (HPI)" was established by the Edwards Lifescience Company (Irvine, California, USA) and is CE certified. As part of the Edwards Acumen Decision-Support-Software-Suite the HPI is supported by the minimal invasive FloTrac Sensor. The HPI displays the probability of an occurring hypotension. The software was established with the help of 20.000 analyzed patient events. If the upper limit of the HPI is reached, the software is alarming the treating physician 8. At the university hospital of Giessen HPI analyses are used in the daily clinical routine as well as for scientific purposes. Preliminary data of the HPI-I-Trial ("Influence of the Hypotension Prediction Index on the number and duration of intraoperative hypotension in primary hip-endoprothetic replacement", University Hospital of Giessen) included patients, which underwent hip-endoprothetic replacement surgery and revealed that the use of HPI with a goal directed therapy (GDT) protocol compared to standard care significantly reduced the incidence and duration of intraoperative hypotension. Therefore HPI with GDT might reduce the incidence of hypotension related complications in a sicker patient cohort.

The development of modern lung surgery started in the 19th century. Especially in Germany Rudolf Nissen (first pneumonectomy, 1931) and Ferdinand Sauerbruch were the first pioneers of lung surgery. With enhancement and refinement of thoracic anesthesiology (lung separation) and further specialization of surgery, thoracic surgery became a seperate discipline. During thoracic surgery lung separation and isolation with accomplished single-lung ventilation plays a key role in the development of thoracic surgery. Spectrum of indication contains thoracic surgery, procedure- and patient-dependent factors. Usually lung isolation is achieved with a double-lumen tube or a bronchial blocker. Major domain of thoracic surgery is nowadays oncological surgery of lung cancer. With modern imaging lung cancer is detected in early stage, so more operations can be performed. Additional in the last thirty years more and more minimal invasive procedures (VATS) were performed which result in gentle and successful treatment of thoracic surgical patients.

Beside oncological surgeries (which make almost 50% of all procedures in thoracic surgery) plays surgery of inflammable diseases and pulmonary emphysema a major role.

Approximately 182.821 thoracic surgical procedures are performed in Germany, 11.451 in Hessen. At the university clinic institution of Giessen more than 500 procedures are performed per year.

Hypotension Prediction Index The "Hypotension Prediction Index (HPI) "was established by the Edwards Lifescience Company (Irvine, USA) and is CE certified. The HPI displays the probability of an occurring hypotension before its onset and therefore can theoretically prevent episodes of hypotension by guiding earlier therapy. This might improve outcome in certain patient populations by preventing episodes of hypotension 29. A recent paper describes the methodology of this prediction tool 25.

Nephro Check NephroCheck is a point of care urine test that flags two biomarkers that indicate if a critically ill patient is at risk for acute kidney injury (AKI) 15. Currently, serum creatinine is the main test used to detect AKI, but it may take a day or more for serum creatinine levels to accumulate in the blood of a patient with a kidney injury consequently, it may not reflect real time kidney damage or loss of function 16. Results of the NephroCheck test are available within 20 minutes before clinical signs of kidney failure are apparent. The evidence suggests that the NephroCheck test has good sensitivity (89% at the 0.3 cutoff value) for detecting critically ill patients at risk for AKI 17, 18.

The aim of the study is to investigate whether a goal directed treatment according to the Hypotension Prediction Index compared to standard care can reduce the incidence of intraoperative hypotension in patients under single lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung surgery with one-lung-ventilation
* General anesthesia
* Age ≥ 18 years

Exclusion Criteria:

* Participation in another (interventional) study
* Pregnancy and nursing mothers
* Surgery without controlled ventilation
* ASA I or IV
* Contraindication for invasive blood pressure monitoring
* Coagulation disorder
* Arterial Fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | up to 8 hours
  Frequency (n) and duration (t [min]) of intraoperative hypotension, defined as MAP below 65mmHg for one minute.

SECONDARY OUTCOMES:
Renal failure | preoperative, immediately after operation and day 1 after operation
  Acute Kidney Injury Risk Score: (TIMP-2)x(IGFBD-7) The product of the measured concentrations out of a urin sample of the two biomarkers, TIMP-2 and IGFBP-7 (measured as ng/mL), divided by 1000 is the result measured as AKI (AcuteKidneyInjury) Risk score. Based upon results from clinical testing, intended use patients with AKIRISK® Scores < 0.3 are at lower risk of developing moderate to severe AKI within 12 hours of assessment than intended use patients with AKIRISK® Scores > 0.3.
Concentration of troponin | preoperative, immediately after operation and day 1 after operation
  MINS (Myocardiac injury after non-cardiac injury) defined as high troponin (µg/l) levels after admission to the ICU and day 1 after surgery
Hemodynamic status | up to 8 hours
  Volume loss and intake of iv fluids (crystalloid, colloidal, blood products and autologous blood) (in ml)
Procedual Data | until the end of anesthesia
  Duration of surgery and anesthesia
POMS (Postoperative Morbidity Survey Score) | day 1, 3 and 5 after operation
  Postoperative Morbidity Survey Score. This score evaluates morbidity after elective surgery monitoring nine different categories.
Circulation supportive mediaction | from beginning until the end of surgery
  Type and dosage of vasopressors and inotropic medication used during the procedure (in µg)
Hospital stay | From admission to hospital until discharge of hospital up to 18 month
  Hospital length of stay (in minutes) and Intensive care (ICU and IMCU) length of stay (in minutes)
Mortality after surgery | up to 180 days after surgery
  Survival postoperative, 90 days after surgery, 180 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, Prof., Study Chair — Study Chair, Head of Department
Locations (1):
- Univeristy of Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007 Aug;107(2):213-20. doi: 10.1097/01.anes.0000270724.40897.8e. PMID 17667564
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] van Waes JA, van Klei WA, Wijeysundera DN, van Wolfswinkel L, Lindsay TF, Beattie WS. Association between Intraoperative Hypotension and Myocardial Injury after Vascular Surgery. Anesthesiology. 2016 Jan;124(1):35-44. doi: 10.1097/ALN.0000000000000922. PMID 26540148
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Morris RW, Watterson LM, Westhorpe RN, Webb RK. Crisis management during anaesthesia: hypotension. Qual Saf Health Care. 2005 Jun;14(3):e11. doi: 10.1136/qshc.2002.004440. PMID 15933284
- [Background] Reich DL, Hossain S, Krol M, Baez B, Patel P, Bernstein A, Bodian CA. Predictors of hypotension after induction of general anesthesia. Anesth Analg. 2005 Sep;101(3):622-628. doi: 10.1213/01.ANE.0000175214.38450.91. PMID 16115962
- [Background] de Mendonca A, Vincent JL, Suter PM, Moreno R, Dearden NM, Antonelli M, Takala J, Sprung C, Cantraine F. Acute renal failure in the ICU: risk factors and outcome evaluated by the SOFA score. Intensive Care Med. 2000 Jul;26(7):915-21. doi: 10.1007/s001340051281. PMID 10990106
- [Background] Liu YL, Prowle J, Licari E, Uchino S, Bellomo R. Changes in blood pressure before the development of nosocomial acute kidney injury. Nephrol Dial Transplant. 2009 Feb;24(2):504-11. doi: 10.1093/ndt/gfn490. Epub 2008 Sep 3. PMID 18768582
- [Background] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Background] Owens P, O'Brien E. Hypotension in patients with coronary disease: can profound hypotensive events cause myocardial ischaemic events? Heart. 1999 Oct;82(4):477-81. doi: 10.1136/hrt.82.4.477. PMID 10490564
- [Background] Mitchinson MJ. The hypotensive stroke. Lancet. 1980 Feb 2;1(8162):244-6. doi: 10.1016/s0140-6736(80)90728-x. PMID 6101689
- [Background] Ovbiagele B, Diener HC, Yusuf S, Martin RH, Cotton D, Vinisko R, Donnan GA, Bath PM; PROFESS Investigators. Level of systolic blood pressure within the normal range and risk of recurrent stroke. JAMA. 2011 Nov 16;306(19):2137-44. doi: 10.1001/jama.2011.1650. PMID 22089721
- [Background] Merx H, Dreinhofer K, Schrader P, Sturmer T, Puhl W, Gunther KP, Brenner H. International variation in hip replacement rates. Ann Rheum Dis. 2003 Mar;62(3):222-6. doi: 10.1136/ard.62.3.222. PMID 12594106
- [Background] Kam Tao Li P, Burdmann EA, Mehta RL; World Kidney Day Steering Committee 2013. Acute kidney injury: Global health alert. J Nephropathol. 2013 Apr;2(2):90-7. doi: 10.12860/JNP.2013.15. Epub 2013 Apr 1. PMID 24475433
- [Background] Lewington AJ, Sayed A. Acute kidney injury: how do we define it? Ann Clin Biochem. 2010 Jan;47(Pt 1):4-7. doi: 10.1258/acb.2009.009249. PMID 20040796
- [Background] Martensson J, Martling CR, Bell M. Novel biomarkers of acute kidney injury and failure: clinical applicability. Br J Anaesth. 2012 Dec;109(6):843-50. doi: 10.1093/bja/aes357. Epub 2012 Oct 9. PMID 23048068
- [Background] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Background] Kashani K, Al-Khafaji A, Ardiles T, Artigas A, Bagshaw SM, Bell M, Bihorac A, Birkhahn R, Cely CM, Chawla LS, Davison DL, Feldkamp T, Forni LG, Gong MN, Gunnerson KJ, Haase M, Hackett J, Honore PM, Hoste EA, Joannes-Boyau O, Joannidis M, Kim P, Koyner JL, Laskowitz DT, Lissauer ME, Marx G, McCullough PA, Mullaney S, Ostermann M, Rimmele T, Shapiro NI, Shaw AD, Shi J, Sprague AM, Vincent JL, Vinsonneau C, Wagner L, Walker MG, Wilkerson RG, Zacharowski K, Kellum JA. Discovery and validation of cell cycle arrest biomarkers in human acute kidney injury. Crit Care. 2013 Feb 6;17(1):R25. doi: 10.1186/cc12503. PMID 23388612
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Mascha EJ, Yang D, Weiss S, Sessler DI. Intraoperative Mean Arterial Pressure Variability and 30-day Mortality in Patients Having Noncardiac Surgery. Anesthesiology. 2015 Jul;123(1):79-91. doi: 10.1097/ALN.0000000000000686. PMID 25929547
- [Background] Vernooij LM, van Klei WA, Machina M, Pasma W, Beattie WS, Peelen LM. Different methods of modelling intraoperative hypotension and their association with postoperative complications in patients undergoing non-cardiac surgery. Br J Anaesth. 2018 May;120(5):1080-1089. doi: 10.1016/j.bja.2018.01.033. Epub 2018 Mar 21. PMID 29661385
- [Background] Sessler DI, Khanna AK. Perioperative myocardial injury and the contribution of hypotension. Intensive Care Med. 2018 Jun;44(6):811-822. doi: 10.1007/s00134-018-5224-7. Epub 2018 Jun 4. PMID 29868971
- [Background] Devereaux PJ, Duceppe E, Guyatt G, Tandon V, Rodseth R, Biccard BM, Xavier D, Szczeklik W, Meyhoff CS, Vincent J, Franzosi MG, Srinathan SK, Erb J, Magloire P, Neary J, Rao M, Rahate PV, Chaudhry NK, Mayosi B, de Nadal M, Iglesias PP, Berwanger O, Villar JC, Botto F, Eikelboom JW, Sessler DI, Kearon C, Pettit S, Sharma M, Connolly SJ, Bangdiwala SI, Rao-Melacini P, Hoeft A, Yusuf S; MANAGE Investigators. Dabigatran in patients with myocardial injury after non-cardiac surgery (MANAGE): an international, randomised, placebo-controlled trial. Lancet. 2018 Jun 9;391(10137):2325-2334. doi: 10.1016/S0140-6736(18)30832-8. PMID 29900874
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Joosten A, Coeckelenbergh S, Delaporte A, Ickx B, Closset J, Roumeguere T, Barvais L, Van Obbergh L, Cannesson M, Rinehart J, Van der Linden P. Implementation of closed-loop-assisted intra-operative goal-directed fluid therapy during major abdominal surgery: A case-control study with propensity matching. Eur J Anaesthesiol. 2018 Sep;35(9):650-658. doi: 10.1097/EJA.0000000000000827. PMID 29750699
- See also: American Society of Anesthesiologists — https://education.asahq.org/totara/course/view.php?id=2947
- See also: EDWARDS HPI — https://www.edwards.com/de/devices/decision-software/hpi